CLINICAL TRIAL: NCT00316732
Title: Observational Sutdy to Assess the Effectiveness of Avodart in Subjects With Benign Prostatic Hyperplasia in Day to Day Clinical Practice
Brief Title: Observational AVODART (Dutasteride) Study In Benign Prostatic Hyperplasia Subjects - OASIS
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 103500
Record Dates: First submitted 2006-04-20; First posted 2006-04-21 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Prostatic Hyperplasia
Keywords: Avodart; IPSS; BPH; dutasteride; EQ-5D; Observational
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: IPSS Questionnaire
Procedure: EQ-5D Questionnaire
  Other Names: IPSS Questionnaire

SUMMARY:
This study was designed to assess the effectiveness of dutasteride in the actual clinical practice of prostate assessment clinics in the UK in accordance with best practice over a 12-month period.

ELIGIBILITY:
Inclusion Criteria:

* Patients who not have received any pharmacological treatment or surgical interventions for BPH (Benign Prostatic Hyperplasia).
* Patients should be prescribed dutasteride in compliance with the UK SmPC and BAUS guidelines on the treatment of BPH.
* Patients must only enter the study after the decision to prescribe dutasteride has been undertaken.

Exclusion criteria: None specified

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2004-10-25 (Actual); Primary Completion 2006-12-19 (Actual); Study Completion 2006-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (23):
- United Kingdom (23):
  - GSK Investigational Site, Exeter, Devon
  - GSK Investigational Site, Plymouth, Devon
  - GSK Investigational Site, Colchester, Essex
  - GSK Investigational Site, Stevenage, Hertfordshire
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, Leicester, Leicestershire
  - GSK Investigational Site, Leytonstone, London
  - GSK Investigational Site, Enfield, Middlesex
  - GSK Investigational Site, Nottingham, Nottinghamshire
  - GSK Investigational Site, Tauton, Somerset
  - GSK Investigational Site, Sunderland, Tyne & Wear
  - GSK Investigational Site, Sutton Coldfield, West Midlands
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, East Kilbride
  - GSK Investigational Site, Hull
  - GSK Investigational Site, Ilkeston, Derbyshire
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, London
  - GSK Investigational Site, Sheffield
  - GSK Investigational Site, Torquay
  - GSK Investigational Site, Wakefield